CLINICAL TRIAL: NCT00746512
Title: A Randomized, Double-Blind, Parallel Group, Placebo Controlled Study to Access the Effects of Oral Prednisone on Clinical Efficacy and the Power Doppler Ultrasound Signal of Synovium in Patients With Rheumatoid Arthritis
Brief Title: A Study of the Effects of Oral Prednisone in Patients With Rheumatoid Arthritis (MK0000-088)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-088; 2008_531
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Results first posted 2011-04-08 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Prednisone 15 mg (Experimental): Prednisone 15 mg tablets once daily for 15 days
  Interventions: Drug: Prednisone 15 mg
- Placebo 15 mg (Placebo Comparator): Prednisone 15 mg placebo tablets once daily for 15 days
  Interventions: Drug: Placebo Tablets
- Prednisone 7.5 mg (Experimental): Prednisone 7.5 mg over-encapsulated tablets once daily for 15 days
  As per adaptive dose-ranging design, this arm was added to the study because a difference between prednisone 15 mg and placebo was demonstrated during interim analysis.
  Interventions: Drug: Prednisone 7.5 mg
- Placebo 7.5 mg (Placebo Comparator): Prednisone 7.5 mg placebo over-encapsulated tablets once daily for 15 days
  As per adaptive dose-ranging design, this arm was added to the study because a difference between prednisone 15 mg and placebo was demonstrated during interim analysis.
  Interventions: Drug: Placebo Over-Encapsulated Tablets

INTERVENTIONS:
Drug: Prednisone 15 mg — Prednisone 15 mg tablets once daily for 15 days.
  Other Names: Prednisone
  Arms: Prednisone 15 mg
Drug: Placebo Tablets — Prednisone placebo tablets once daily for 15 days.
  Arms: Placebo 15 mg
Drug: Prednisone 7.5 mg — Prednisone 7.5 mg over-encapsulated tablets once daily for 15 days
  Other Names: Prednisone
  Arms: Prednisone 7.5 mg
Drug: Placebo Over-Encapsulated Tablets — Prednisone 7.5 mg placebo over-encapsulated tablets once daily for 15 days
  Arms: Placebo 7.5 mg

SUMMARY:
The study will compare the effects of prednisone vs placebo on synovial blood flow and overall DAS (disease activity score) in patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing to limit alcohol intake to 3 or less beverages per day
* Patient agrees to use only acetaminophen/paracetamol for breakthrough pain

Exclusion Criteria:

* Patient has other inflammatory arthritis (e.g. lupus). Patient has had major surgery or donated or lost 1 unit of blood in the last 4 weeks
* Patient has a history of drug or alcohol abuse in the last 2 years
* Patient has had a vaccine (with a live or attenuated virus) in the last two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Seymour MW, Kelly S, Beals CR, Malice MP, Bolognese JA, Dardzinski BJ, Cheng AS, Cummings CE, Smugar SS, McClinton C, Fox A, Dooley WM, Pitzalis C, Taylor PC. Ultrasound of metacarpophalangeal joints is a sensitive and reliable endpoint for drug therapies in rheumatoid arthritis: results of a randomized, two-center placebo-controlled study. Arthritis Res Ther. 2012 Sep 12;14(5):R198. doi: 10.1186/ar4034. PMID 22972032

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prednisone 15 mg | Placebo 15 mg | Prednisone 7.5 mg | Placebo 7.5 mg
Started | 8 | 10 | 18 | 9
Completed | 8 | 10 | 18 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prednisone 15 mg | Placebo 15 mg | Prednisone 7.5 mg | Placebo 7.5 mg | Total
Number analyzed (Participants) | 8 | 10 | 18 | 9 | 45
Age, Continuous [Mean (Full Range); unit: years] | 61.6 [48 to 69] | 58.4 [45 to 86] | 57.9 [37 to 81] | 55.1 [32 to 71] | 58.1 [32 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 12 | 6 | 29
  Male | 2 | 5 | 6 | 3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Synovial Blood Flow
Description: Synovial Blood Flow was measured as the 2-dimensional quantitative Transverse Power Doppler Area summed over each of the 10 metacarpophalangeal joints (10MCP 2D Trans PDA). The PDA is a count of the number of pixels with power Doppler signal, uncorrected by pixel intensity, within an expert drawn region of interest encompassing the synovium and excluding digital vessels in a standardized 2D transverse image of the joint. A higher pixel count relates to greater synovial blood flow. A decrease in pixel count relates to a reduction in synovial blood flow.
Time Frame: Baseline and Day 14
Measure: Mean (Standard Deviation); unit: pixel count
Arm/Group | Prednisone 15 mg | Placebo 15 mg | Prednisone 7.5 mg | Placebo 7.5 mg
Number analyzed (Participants) | 8 | 10 | 18 | 9
pixel count
  Baseline | 9.48 (6.44) | 10.55 (9.54) | 8.31 (8.66) | 9.78 (7.28)
  Day 14 | 6.52 (6.40) | 13.37 (11.05) | 4.44 (4.94) | 9.15 (11.65)
  Change from Baseline at Day 14 | -2.96 (5.07) | 2.82 (4.62) | -3.88 (5.71) | -0.64 (9.41)

2. Secondary Outcome: Disease Activity Score 28 (DAS28) (C-reactive Protein [CRP])
Description: The DAS28(CRP) is a measure of disease activity with components which include the tender joint count (TJC) & swollen joint count (SJC) (each out of 28 joints counted), a Global Health (GH) index (100 mm visual analog scale [VAS]), and the CRP (in mg/L measured from lab test). The scoring formula was:
  DAS28(CRP) = 0.56*SQR(TJC28) + 0.28*SQR(SJC28) + 0.36*ln(CRP+1) + 0.014*GH(VAS) + 0.96.
  Where SQR is square root and ln is natural log.
  The formula produces a score from 0 to 10: >5.1 means high disease activity; <3.2 means low disease activity, <2.6 is generally considered remission.
Time Frame: Baseline and Day 14
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Prednisone 15 mg | Placebo 15 mg | Prednisone 7.5 mg | Placebo 7.5 mg
Number analyzed (Participants) | 8 | 10 | 18 | 9
score on scale
  Baseline | 5.17 (1.30) | 5.45 (1.65) | 5.31 (1.18) | 5.62 (1.78)
  Day 14 | 3.57 (1.50) | 5.04 (2.09) | 4.57 (1.12) | 5.38 (1.60)
  Change from Baseline at Day 14 | -1.61 (1.69) | -0.41 (0.72) | -0.74 (0.86) | -0.23 (0.83)

ADVERSE EVENTS:
Arm/Group | Prednisone 15 mg | Placebo 15 mg | Prednisone 7.5 mg | Placebo 7.5 mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10 | 0/18 | 1/9
Other Adverse Events (participants affected / at risk) | 3/8 | 4/10 | 6/18 | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prednisone 15 mg (N=8) | Placebo 15 mg (N=10) | Prednisone 7.5 mg (N=18) | Placebo 7.5 mg (N=9)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prednisone 15 mg (N=8) | Placebo 15 mg (N=10) | Prednisone 7.5 mg (N=18) | Placebo 7.5 mg (N=9)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Vulvovaginal Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Arthalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Chronic Obstructive Pumonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.